CLINICAL TRIAL: NCT06316765
Title: A Stylet Use May be Beneficial for Elective and Rescue Intubation of Prematurely Born Infants < 30 Weeks.
Brief Title: A Stylet Use May be Beneficial for Elective and Rescue Intubation of Prematurely Born Infants
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Dunajová Klára, Principal Investigator, Charles University, Czech Republic
Other Study IDs: 118/10
Record Dates: First submitted 2024-03-07; First posted 2024-03-18 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Neonatology
Keywords: Resuscitation; Extremely premature infant; Intubation; Stylet
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- With stylet group: Intubation performed with stylet.
  Interventions: Procedure: Intubation with stylet
- Without stylet group: Intubation performed without stylet.

INTERVENTIONS:
Procedure: Intubation with stylet — The cohort of premature infants was intubated with stylet.
  Groups: With stylet group

SUMMARY:
Contrary to recent findings suggesting that stylets offer no advantage in general infant intubations, this study focuses on their potential benefits for premature infants undergoing elective or rescue intubation in the delivery room. The goal is to compare the safety and efficiency of intubations with or without a stylet.

DETAILED DESCRIPTION:
Recent studies have found that using a stylet does not offer any benefits during intubation across a diverse infant population. The research, however, specifically targets extremely and very premature infants undergoing elective or rescue intubation in the delivery room. A single-center retrospective observational study was conducted to compare the number of intubation attempts, the duration of intubation until successful, and the rate of associated desaturations exceeding 20%. The outcomes were determined through video recordings and statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* intubation in the delivery room

Exclusion Criteria:

* both method used, video record not available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All premature infants born at less than 30 weeks gestation between 2016 and 2022 in the General Faculty Hospital in Prague were eligible for evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome was defined as successful initial intubation attempt. | immediately after procedure
  Successful placement of the endotracheal tube on the first intubation attempt, followed by an increase in heart rate and blood oxygen saturation.

SECONDARY OUTCOMES:
Secondary outcomes was defined as the duration of intubation courses until successful placement of the endotracheal tube. | immediately after procedure
  The duration from the first insertion of the laryngoscope blade to the successful placement of the endotracheal tube, followed by an increase in heart rate and blood oxygen saturation, measured in seconds.

IPD SHARING:
Plan to Share IPD: Undecided